CLINICAL TRIAL: NCT02077751
Title: BioRBC Survival in Adults With Prior Antibody Response to BioRBCs
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: John A Widness (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor-Investigator, John A Widness, Professor, Department of Pediatrics, University of Iowa
Organization: University of Iowa (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 200710747-1; 2P01HL046925-16A1 (NIH)
Record Dates: First submitted 2014-02-27; First posted 2014-03-04 (Estimated); Last update posted 2021-04-29 (Actual); Status verified 2021-04

CONDITIONS: Anemia
MeSH Terms: conditions — Anemia

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Biotin labelled RBCs (Experimental): Subjects receive biotin labelled autologous red blood cells.
  Interventions: Drug: biotin labelled RBCs

INTERVENTIONS:
Drug: biotin labelled RBCs — Autologous red blood cells are biotin labelled and transfused to the subject. Survival of these red blood cells is tracked through examination of blood samples until no biotin labelled red blood cells remain.
  Other Names: biotinylated RBCs

SUMMARY:
Objective: To gather safety and efficacy BioRBC data from adult subjects who previously developed transient BioRBC antibody responses by redosing them and observing for adverse clinical or laboratory (i.e., a positive BioRBC antibody titer) outcomes to determine if RBC kinetic study results differ from the previous study.

Hypothesis: BioRBC survival studies performed in adult subjects who previously developed a transient BioRBC antibody response will: 1) be associated with no adverse clinical or laboratory events; 2) experience a second transient, BioRBC antibody response; and 3) display a pattern of RBC survival that is identical to their prior dosing with BioRBCs at the same dose.

DETAILED DESCRIPTION:
Summary. Subjects eligible for study include adult study subjects older than 18 years who had a positive antibody response to BioRBCs in previous BioRBC studies at the University of Iowa, Adult BioRBC Redosing Safety Protocol Page 3 of 6 but who are now BioRBC antibody sero-negative. The study will begin after IRB approval. The information summaries and IRB consent forms used in prior studies did not include a statement indicating that subjects would not be re-contacted for future research. Written informed consent will be obtained prior to study. The total number of subjects available for study is 4, i.e., all subjects who we previously identified as having formed antibodies to BioRBC following autologous BioRBC transfusion.

Removal of subjects. Subjects will be free to withdraw from the study at their discretion. The investigators will also be free to withdraw study subjects from the study for reasons of non-compliance, inability to conduct the required study assessments or if the Investigators determined it was in the best interest of the subject. The reasons for subject withdrawal will be documented. The Investigators will attempt to collect safety data on withdrawn subjects.

Study design. This is an open Phase 1 study in which the only 4 subjects we identified as having developed antibodies to BioRBCs - and who are now negative for these antibodies - will be re-dosed with BioRBCs. This will be conducted at a single study site at the University of Iowa.

As illustrated in the protocol diagram figure below, following screening and enrolment, each subject will donate 100 mL of whole blood collected in CPD preservative from which RBC concentrates will be prepared according to the standard methodology and procedures included in our original 2006 FDA IND application with only minor modification of study sample times.

Specific Aims. Using a dose of biotin labeled autologous RBCs that is ~30% of our previous dose we will determine during a 20 wk post-transfusion study period whether study subjects:

1. Develop a second BioRBC antibody response that is greater than, less than, or equal to each subject's previous response.
2. Experience a fall in Hb/Hct, rise in reticulocyte count, and/or a decrease in RBC survival following the appearance of BioRBC antibodies;
3. Experience clinical signs or symptoms following the appearance of BioRBC antibodies.
4. Have detectable BioRBC enrichment throughout the entire study period (as was possible previously with a larger BioRBC dose).

Dose and duration. A single dose of BioRBCs that will include the same densities of biotin labeled RBCs as studied previously in survival studies. On the first day of study, a fresh ~100 mL aliquot of autologous RBC will be collected and labeled with biotin at densities 6, 18, 54 and 128 μg/mL RBC. Immediately after preparing the four populations of BioRBC densities, the four densities will be combined, mixed, and a gravimetrically determined weight of the blood infused intravenously. An aliquot of the infusate will be saved and analyzed to determine the dose of each density administered.

All labeling will be conducted using approved sterile instruments and materials in a certified laminar flow containment hood to minimize the potential for bacterial contamination. Two aliquots of the BioRBC infusate will be saved: 1) one for endotoxin testing should the subject Adult BioRBC Redosing Safety Protocol Page 5 of 6 develop a transfusion reaction (we have not encountered this in the ~35 adult subjects we have studied to date); and 2) the other for aerobic bacteria cultured for any potential contamination during the labeling process. Although the culture results will not be available prior to the infusion, they will be available in the event the subject develops symptoms of bacterial infection, e.g., fever.

ELIGIBILITY:
Inclusion Criteria:

* Female and male subjects
* Age 18 years or older
* Normal with respect to serum chemistry, and hematology panels. Values outside the normal range, but not considered to be a health risk by the investigator will not exclude a subject
* Consented for the study and have signed an IRB-approved Informed Consent

Exclusion Criteria:

Subjects who had any of the following criteria were excluded from the study:

* History of a clinically significant acute or chronic disease process
* Evidence of previous or current significant cardiovascular (including uncontrolled hypertension), hematologic, gastrointestinal (including hepatic), renal, metabolic, or neurological disorders or clinically significant allergies
* History of autoimmune haemolytic anemia, RBC autoantibodies or alloantibodies, or autoimmune disease
* History of congenital red cell disorders including glucose-6-phosphate dehydrogenase (G-6PD) deficiency
* Positive pregnancy test result
* Whole blood donation within 8 weeks or 2-unit RBC collection within 16 weeks of planned study whole blood donation
* Inability of subject to comply with the protocol in the Investigator's opinion.
* A female who was breast-feeding an infant or child
* Positive Direct or Indirect Antiglobulin Test result
* Immunosuppressive therapy (e.g., oral or intravenous prednisone) within the preceding 28 days
* Subjects who participated in another clinical study concurrently or within 28 days prior to starting the study
* Presence of plasma or serum anti-biotin antibodies to biotinylated RBCs (i.e., RBC labelled at a density of 54 μg/mL when tested using IgG gel card method)

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2013-05 (Actual); Primary Completion 2019-06 (Actual); Study Completion 2019-12 (Actual)

PRIMARY OUTCOMES:
Presence of biotin antibody in blood sample after transfusion of biotinylated RBCs | 10 min to day when antibody is no longer detected, typically 6 months.

CONTACTS AND LOCATIONS:
Overall Officials: John A Widness, MD, Principal Investigator — University of Iowa
Locations (1):
- University of Iowa, Iowa City, Iowa, United States

IPD SHARING:
Plan to Share IPD: No